CLINICAL TRIAL: NCT06758544
Title: A Single-arm, Open-label Clinical Study to Evaluate the Efficacy and Safety of VRT106 in Combination With Chemotherapy for Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Guangzhou Virotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRT106-C05
Record Dates: First submitted 2025-01-02; First posted 2025-01-03 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
Keywords: Resectable pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VRT106 combination with chemotherapy (Experimental): VRT106 combination with chemotherapy
  Interventions: Drug: Oncolytic virus VRT106; Drug: Chemotherapy

INTERVENTIONS:
Drug: Oncolytic virus VRT106 — VRT106, IV
Drug: Chemotherapy — 21 days/cycle, administered up to 6 cycles

SUMMARY:
This is a single-center, single-arm, open investigator-initiated clinical study to evaluate the efficacy and safety of VRT106 in combination with chemotherapy in the treatment of resectable pancreatic cancer.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open investigator-initiated clinical study to evaluate the efficacy and safety of VRT106 in combination with chemotherapy in the treatment of resectable pancreatic cancer.

The study is planned to enroll 18 subjects. The entire study consists of a screening period of up to 28 days, treatment period, and a follow-up period (safety follow-up 28 days after the final study dose and survival follow-up once every 3 months).

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an Institutional Review Board -approved informed consent prior to performing any of the Screening Visit procedures.
2. Males and females at 18-75 years of age, inclusive, at the Screening Visit.
3. Have a clinical diagnosis of pancreatic cancer.
4. An Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
5. Expected survival time of≥6 months.
6. No serious hematologic and cardiac abnormalities of the liver, kidneys, or coagulation functions.

Exclusion Criteria:

1. Prior treatment with other oncolytic virus or systemic therapy for pancreatic cancer.
2. Previous allogeneic hematopoietic stem cell transplantation or organ transplantation.
3. Immunocompromised patients.
4. Known alcohol or drug dependency.
5. Women who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | About 3 years
  Incidence rate of TRAE（Treatment-Related Adverse Event）

SECONDARY OUTCOMES:
Disease-free survival rate | About 2 years
  Disease-free survival rates at 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No